CLINICAL TRIAL: NCT05260645
Title: Prevention of Neck Pain in Adults With a Back School-Based Intervention.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5148
Record Dates: First submitted 2022-02-08; First posted 2022-03-02 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Neck Pain; Exercise Therapy; Health Education; Primary Prevention
MeSH Terms: conditions — Neck Pain; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Intervention based on the Back School was carried out for 8 weeks with a frequency of two sessions per week, with a total of 16 sessions lasting 45 min.
  Interventions: Behavioral: Back School
- Control group (No Intervention): I declare that I will not change my lifestyle during the study process.

INTERVENTIONS:
Behavioral: Back School — Intervention was carried out for 8 weeks with a frequency of two sessions per week, with a total of 16 sessions lasting 45 min. Of all the sessions, 14 had a practical focus and the other two had a theoretical focus. In the practical part, strengthening and stretching exercises were performed. In the theoretical part, self-management and pain neuroscience education were performed.
  Arms: Experimental group

SUMMARY:
The study consists of a theoretical and practical intervention based on the Back School. This intervention will be carried out over 8 weeks with a frequency of two sessions per week, for a total of 16 sessions of 45 minutes duration. Of all the sessions, 14 had a practical focus (strength and stretching exercises) and the other two had a theoretical focus (self-management techniques and pain neuroscience education).

The clinical practice guidelines highlight the importance of neck pain prevention through exercise an education. There are previous studies of the effects of theoretical and practical programmes based on back school on the lumbar region but not on the cervical region.Therefore, the main aim of this innovative study is to to investigate the effects of a Back School based intervention on the prevention of neck pain and as secondary objectives to investigate the effects on neck flexor and extensor strength as well as scapular stability. The hypothesis is that this BS-based intervention would have positive effects on neck pain prevention, neck strength and scapular stability.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 65 years old.
* Not have had neck pain in the last 6 months.

Exclusion Criteria:

* Previous neck or shoulder surgery, cervical radiculopathy/myelopathy, history of the whiplash injury.
* Taking any medication or having any musculoskeletal, rheumatic, metabolic, cardiological, cognitive disorder or neurological disorder.
* Missing more than two Back School sessions.
* Not being able to attend the measurement sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Changes in the incidence of neck pain. | From the end of the back school intervention until 12 months of follow-up
  Participants recorded the number of episodes of neck pain in a diary.
Changes in the duration of neck pain. | From the end of the back school intervention until 12 months of follow-up
  Participants recorded the number of days of neck pain in a diary.
Changes in the Numeric Pain Rating Scale. | From the end of the back school intervention until 12 months of follow-up
  Participants recorded neck pain intensity in a diary using the Numeric Pain Rating Scale (0-10). The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Changes in the medical visits from baseline to eight months. | From the end of the back school intervention until 12 months of follow-up
  Participants recorded the number of medical visits for neck pain in a diary. These data were collected at the end of the intervention and at 6-month follow-up.

SECONDARY OUTCOMES:
Neck flexor muscle endurance. | Baseline and two months.
  This was measured using the deep neck flexor endurance test as described by Grimmer (1994). When in supine position, participants were asked to flex the upper cervical spine, move their heads away from the couch approximately 2.5 cm and hold this position for as long as possible. The test ended when students dropped their heads or lost craniocervical flexion.
Neck extensor muscle endurance. | Baseline and two months.
  The neck extensor endurance test was performed in line with the guidelines by Edmondston et al (2008). Students were in prone position, head neutral, arms by their sides and a 10-cm stabilising strip of Velcro was placed at the sixth dorsal vertebra level. An inclinometer and 5-cm strap were placed around the participants head with a 2-kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining a neutral head position.
Scapular stabiliser endurance | Baseline and two months.
  Endurance of the scapular stabilisers was assessed as described by Edmondston et al (2008). Participants stood with their shoulders and elbows flexed at 90°. Students' elbows were kept approximately shoulder-distance apart with a ruler and they were asked to pull both extremities of the dynamometer by externally rotating their shoulders until the dynamometer reached 1 kg. They were asked to hold this position for as long as possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Pablo Hernández Lucas, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hernandez-Lucas P, Leiros-Rodriguez R, Lopez-Barreiro J, Garcia-Soidan JL. Prevention of neck pain in adults with a Back School-Based intervention: a randomized controlled trial. Physiother Theory Pract. 2025 Jan;41(1):54-64. doi: 10.1080/09593985.2024.2316313. Epub 2024 Feb 16. PMID 38362871